CLINICAL TRIAL: NCT02191878
Title: Open-Label, Multi-Center, Phase 1, Dose Escalation Study With Phase 2 Expansion Cohort to Determine the Safety, Pharmacokinetics and Preliminary Anti-Tumor Activity of Intravenous TKM-080301 in Subjects With Advanced Hepatocellular Carcinoma
Brief Title: Safety, Pharmacokinetics and Preliminary Anti-Tumor Activity of Intravenous TKM-080301 in Subjects With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arbutus Biopharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TKM-HCC-001
Record Dates: First submitted 2014-07-09; First posted 2014-07-16 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Hepatocellular Carcinoma; Hepatoma; Liver Cancer, Adult; Liver Cell Carcinoma, Adult
Keywords: Liver Cancer; Liver Neoplasms; Liver Epithelial Neoplasms; Liver Cancer, malignant
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — TKM-080301

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase 1 Escalation / Phase 2 Expansion (Experimental): Phase 1 - dose escalation with intravenous infusion of TKM-080301 to determine MTD.
  Phase 2 - dose expansion at the MTD.
  Interventions: Drug: TKM-080301

INTERVENTIONS:
Drug: TKM-080301 — TKM-080301 intravenous infusion
  Other Names: PLK1-HCC

SUMMARY:
This study is an open-label, multi-center, phase 1, dose escalation study with a phase 2 expansion cohort to determine the safety, pharmacokinetics and preliminary anti-tumor activity of intravenous TKM-080301 in subjects with advanced hepatocellular carcinoma (HCC).

This study is being done to:

* Test the safety and tolerability of TKM-080301 in subjects with advanced hepatocellular carcinoma
* Find the highest dose of TKM-080301 that can be given without causing side effects, called the maximum tolerated dose (MTD).
* Provide a preliminary assessment of anti-tumor activity of TKM-080301

DETAILED DESCRIPTION:
Study design: Open label, multi-center, 3 + 3 dose-escalation study with an expansion cohort at the maximum tolerated dose (MTD) to investigate safety, tolerability, PK, and preliminary anti-tumor activity of TKM 080301 in subjects with HCC.

Sequential cohorts of 3 to 6 subjects will receive escalating doses of TKM 080301 according to a pre-specified dose escalation scheme. Assessment of dose-limiting toxicities (DLTs) will be made during Cycle 1 to determine the maximum tolerated dose (MTD). Once the MTD level is established, approximately 20 subjects will be enrolled in an expansion cohort to further confirm the safety and tolerability of TKM-080301 at the MTD.

Study Population: A minimum of 9 and up to approximately 18 adult male or female subjects with histologically or cytologically confirmed metastatic or locally advanced inoperable HCC and a life expectancy of 3 months or more are planned in the dose escalation phase. Approximately 20 subjects are planned in the expansion cohort.

Study Treatment: TKM-080301 will be administered by intravenous (IV) infusion, once weekly for 3 consecutive weeks followed by a 1 week rest period. This 28-day treatment period constitutes 1 cycle.

Subjects who demonstrate clinical benefit without progression per RECIST 1.1 guidelines may receive treatment beyond 6 cycles if the Investigator considers it is in the best interest of the subject, and only with the approval of the Medical Monitor. Subjects would then continue TKM 080301 therapy until withdrawal of consent, disease progression or unacceptable toxicity occurs.

Pharmacokinetics (PK) Subjects will undergo blood sample collection for PK analysis during cycles 1 and 2.

Study Duration: Each treatment cycle will have duration of 28 days and each subject will typically receive up to 6 cycles of treatment. The total duration of the study is expected to be approximately 28 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Child-Pugh class of A
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5.0 × ULN
* Total bilirubin ≤3.0 mg/dL
* Platelets ≥75,000 /mL
* International Normalized Ratio (INR) ≤1.7
* Subjects must meet the protocol-defined criteria for both hepatitis B virus (HBV) and hepatitis C virus (HCV) status

Key Exclusion Criteria:

* History of significant cardiovascular disease will be excluded
* History of liver transplant.
* Diagnosis of fibrolamellar HCC or tumors of mixed histology.
* Subjects known to be positive for Human immunodeficiency virus (HIV) infection.
* Known central nervous system (CNS) or brain metastases.
* Poorly controlled ascites and/or requirement for therapeutic paracentesis more frequently than once every 3 months.
* Symptomatic encephalopathy within 3 months prior to the first dose of TKM-080301 and/or requirement for medication for encephalopathy.
* Esophageal variceal bleeding within 2 weeks prior to the first dose of TKM-080301.
* Asthma or chronic obstructive pulmonary disease (COPD) requiring daily medication.
* Prior therapy with nitrosoureas or mitomycin within 6 weeks prior to the first dose of TKM-080301.
* Prior therapy with any biologic chemotherapeutic or investigational drug within 5 half-lives or 3 weeks, whichever is longer prior to the first dose of TKM 080301.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 6 months after initial dose.
  Laboratory assessments

SECONDARY OUTCOMES:
Preliminary assessment of anti-tumor activity by Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1) | Upon every 2 cycles of treatment for up to 6 months
  Obtain preliminary assessment of anti-tumor activity by Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1)
Clinical Benefit Rate at maximum tolerated dose (MTD) in Expansion Cohort | Upon completion of treatment of expansion cohort; up to 6 months after last participant is dosed.
  Assessed after completion of Phase 2.

OTHER OUTCOMES:
Assessment of Pharmacodynamic Effect | Upon completion of cycle 1 and cycle 2 treatment; 1 and 2 months after last participant is dosed in expansion cohort.
  Assessment of target mRNA reduction in participants consenting to pre- and post-treatment tumor biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kowalski, M.D., Ph.D., Study Director — Tekmira Pharmaceuticals
Locations (15):
- United States (5):
  - Arizona Clinical Research Center, Tucson, Arizona
  - University of California San Francisco, San Francisco, California
  - Kansas City Research Institute, Kansas City, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Mary Crowley Cancer Research Centers, Dallas, Texas
- Princess Margaret Hospital, Toronto, Ontario, Canada
- Queen Mary Hospital, Hong Kong, China
- National University Hospital, Singapore, Singapore
- South Korea (4):
  - Seoul National University Hospital, Seoul, Gyeonggi-do
  - Samsung Medical Center, Seoul, Gyeonggi-do
  - ASAN Medical Center, Seoul, Gyeonggi-do
  - Severence Hospital, Yonsei, University Health System, Seoul
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Shuang-Ho Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Derived] El Dika I, Lim HY, Yong WP, Lin CC, Yoon JH, Modiano M, Freilich B, Choi HJ, Chao TY, Kelley RK, Brown J, Knox J, Ryoo BY, Yau T, Abou-Alfa GK. An Open-Label, Multicenter, Phase I, Dose Escalation Study with Phase II Expansion Cohort to Determine the Safety, Pharmacokinetics, and Preliminary Antitumor Activity of Intravenous TKM-080301 in Subjects with Advanced Hepatocellular Carcinoma. Oncologist. 2019 Jun;24(6):747-e218. doi: 10.1634/theoncologist.2018-0838. Epub 2018 Dec 31. PMID 30598500